CLINICAL TRIAL: NCT02940262
Title: 68Ga-PSMA PET/CT for Detection of Recurrent Prostate Cancer After Initial Therapy
Brief Title: Gallium Ga 68-labeled PSMA-11 PET/CT in Detecting Recurrent Prostate Cancer in Patients After Initial Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-001095; NCI-2016-01212 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-10-19; First posted 2016-10-20 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Prostate Adenocarcinoma; Recurrent Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (68Ga-PSMA-11) (Experimental): Patients receive gallium Ga 68-labeled PSMA-11 IV. Beginning 50-100 minutes after receiving gallium Ga 68-labeled PSMA-11, patients undergo PET imaging.
  Interventions: Radiation: Gallium Ga 68 Gozetotide; Other: Laboratory Biomarker Analysis; Procedure: Positron Emission Tomography

INTERVENTIONS:
Radiation: Gallium Ga 68 Gozetotide — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; Gallium Ga 68 PSMA-11; Gallium Ga 68-labeled PSMA-11; GALLIUM GA-68 GOZETOTIDE; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Positron Emission Tomography — Undergo PET imaging
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This clinical trial studies how well gallium Ga 68-labeled prostate-specific membrane antigen (PSMA)-11 positron emission tomography (PET)/computed tomography (CT) works in detecting prostate cancer that has come back (recurrent) in patients after initial therapy. Diagnostic procedures, such as gallium Ga 68-labeled PSMA-11 PET/CT, may help doctors detect tumors that have come back after initial therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the sensitivity on a per-patient and per-region-basis of Gallium Ga 68 Gozetotide (68Ga-PSMA-11) PET for detection of tumor location confirmed by histopathology/biopsy, clinical and conventional imaging follow-up.

SECONDARY OBJECTIVES:

I. To assess the positive predictive value (PPV) on a per-patient and per-region-basis of 68Ga-PSMA-11 PET for detection of tumor location confirmed by histopathology/biopsy, clinical and conventional imaging follow-up (composite reference standard).

II. To assess the sensitivity and positive predictive value (PPV) on a per-patient and per-region-basis of 68Ga-PSMA-11 PET for detection of tumor location confirmed by histopathology/biopsy only.

III. To assess the detection rates on a per-patient basis of 68Ga-PSMA-11 PET stratified by prostate specific antigen (PSA) value (0.2 - < 0.5, 0.5 - < 1.0, 1.0 - < 2.0, 2.0 - < 5.0, >= 5.0).

IV. To assess the impact of 68Ga-PSMA-11 PET on clinical management in biochemical recurrence (BCR) patients.

V. To assess the inter-reader reproducibility. VI. To assess the safety of 68Ga-PSMA-11 PET. VII. To assess the detection rates on a per-patient basis of 68Ga-PSMA-11 PET stratified by PSA velocity and PSA doubling-time.

OUTLINE:

Patients receive gallium Ga 68-labeled PSMA-11 intravenously (IV). Beginning 50-100 minutes after receiving gallium Ga 68-labeled PSMA-11, patients undergo PET imaging.

After completion of study, patients are followed up for 3-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological proven prostate adenocarcinoma
* Rising PSA after definitive therapy with prostatectomy or radiation therapy.

  * Post radical prostatectomy (RP)

    * PSA equals to or greater than 0.2 ng/mL measured more than 6 weeks after RP
  * Post-radiation therapy - American Society for Therapeutic Radiation and Oncology (ASTRO)-Phoenix consensus definition

    * Nadir + greater than or equal to 2 ng/mL rise in PSA
* Karnofsky performance status of >= 50 (or Eastern Cooperative Oncology Group [ECOG]/ World Health Organization [WHO] equivalent)
* Ability to understand a written informed consent document, and the willingness to sign it

Exclusion Criteria:

* Concomitant investigational therapy
* Known inability to lie flat, remain still or tolerate a PET scan
* Patient undergoing active treatment for non-prostate malignancy, other than skin basal cell or cutaneous superficial squamous cell carcinoma that has not metastasized and superficial bladder cancer

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1138 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Sensitivity on a per-patient and per-region-basis of gallium Ga 68-labeled PSMA-11 positron emission tomography for detection of tumor location | Up to 12 months
  Confirmed by histopathology/biopsy, clinical and conventional imaging follow-up. Will be calculated and reported along with the corresponding two-sided 95% confidence intervals. The confidence intervals will be constructed using the Wilson score method.

SECONDARY OUTCOMES:
Positive predictive value (PPV) on a per-patient and per-region-basis of gallium Ga 68-labeled PSMA-11 positron emission tomography for detection of tumor location | Up to 12 months
  Confirmed by histopathology/biopsy and, clinical and conventional imaging follow-up. Will be calculated and reported along with the corresponding two-sided 95% confidence intervals. The paired McNemar's test will be used to compare the positive predictive values of gallium Ga 68-labeled PSMA-11 positron emission tomography imaging to the positive predictive values of conventional imaging.
Sensitivity and PPV on a per-patient and per-region-basis of 68Ga-PSMA-11 positron emission tomography (PET) for detection of tumor location confirmed by histopathology/biopsy | Up to 12 months
  Will be summarized in tabular format. Ninety-five confidence intervals of sensitivity, specificity, and net present value (NPV) will be calculated using the Wilson score method.
Detection rates on a per-patient basis of gallium Ga 68-labeled PSMA-11 positron emission tomography stratified by PSA value | Up to 12 months
  Detection rates on a per-patient basis of gallium Ga 68-labeled PSMA-11 positron emission tomography stratified by PSA value (0.2 - < 0.5, 0.5 - < 1.0, 1.0 - < 2.0, 2.0 - < 5.0, >= 5.0) and PSA velocity/doubling-time will be summarized in tabular format and compared between PSA strata using chi-square analysis.
Detection rates on a per-patient basis of gallium Ga 68-labeled PSMA-11 positron emission tomography stratified by PSA velocity and PSA doubling-time | Up to 12 months
  Detection rates on a per-patient basis of gallium Ga 68-labeled PSMA-11 positron emission tomography stratified by PSA value (0.2 - < 0.5, 0.5 - < 1.0, 1.0 - < 2.0, 2.0 - < 5.0, >= 5.0) and PSA velocity/doubling-time will be summarized in tabular format and compared between PSA strata using chi-square analysis.
Clinical management in biochemical recurrence patients | Up to 12 months
  The impact of gallium Ga 68-labeled PSMA-11 positron emission tomography on clinical management in biochemical recurrence patients will be evaluated using descriptive statistics.
Inter-reader reproducibility | Up to 12 months
  Inter-reader reproducibility for positivity at the patient level and region level will be reported using the Fleiss' Kappa test for multiple readers.
Incidence of adverse events | Up to 12 months
  Safety will be reported descriptively as rates of patient reported adverse events. Additionally, adverse events will be characterized and quantified by Common Terminology Criteria for Adverse Events 4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Czernin, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Fendler WP, Calais J, Eiber M, Simko JP, Kurhanewicz J, Santos RD, Feng FY, Reiter RE, Rettig MB, Nickols NG, Kishan AU; PSMA PET Reader Group; Slavik R, Carroll PR, Lawhn-Heath C, Herrmann K, Czernin J, Hope TA. False positive PSMA PET for tumor remnants in the irradiated prostate and other interpretation pitfalls in a prospective multi-center trial. Eur J Nucl Med Mol Imaging. 2021 Feb;48(2):501-508. doi: 10.1007/s00259-020-04945-1. Epub 2020 Aug 17. PMID 32808077
- [Derived] Calais J, Ceci F, Eiber M, Hope TA, Hofman MS, Rischpler C, Bach-Gansmo T, Nanni C, Savir-Baruch B, Elashoff D, Grogan T, Dahlbom M, Slavik R, Gartmann J, Nguyen K, Lok V, Jadvar H, Kishan AU, Rettig MB, Reiter RE, Fendler WP, Czernin J. 18F-fluciclovine PET-CT and 68Ga-PSMA-11 PET-CT in patients with early biochemical recurrence after prostatectomy: a prospective, single-centre, single-arm, comparative imaging trial. Lancet Oncol. 2019 Sep;20(9):1286-1294. doi: 10.1016/S1470-2045(19)30415-2. Epub 2019 Jul 30. PMID 31375469
- [Derived] Fendler WP, Calais J, Eiber M, Flavell RR, Mishoe A, Feng FY, Nguyen HG, Reiter RE, Rettig MB, Okamoto S, Emmett L, Zacho HD, Ilhan H, Wetter A, Rischpler C, Schoder H, Burger IA, Gartmann J, Smith R, Small EJ, Slavik R, Carroll PR, Herrmann K, Czernin J, Hope TA. Assessment of 68Ga-PSMA-11 PET Accuracy in Localizing Recurrent Prostate Cancer: A Prospective Single-Arm Clinical Trial. JAMA Oncol. 2019 Jun 1;5(6):856-863. doi: 10.1001/jamaoncol.2019.0096. PMID 30920593
- [Derived] Calais J, Fendler WP, Herrmann K, Eiber M, Ceci F. Comparison of 68Ga-PSMA-11 and 18F-Fluciclovine PET/CT in a Case Series of 10 Patients with Prostate Cancer Recurrence. J Nucl Med. 2018 May;59(5):789-794. doi: 10.2967/jnumed.117.203257. Epub 2017 Dec 14. PMID 29242404
- [Derived] Calais J, Fendler WP, Eiber M, Gartmann J, Chu FI, Nickols NG, Reiter RE, Rettig MB, Marks LS, Ahlering TE, Huynh LM, Slavik R, Gupta P, Quon A, Allen-Auerbach MS, Czernin J, Herrmann K. Impact of 68Ga-PSMA-11 PET/CT on the Management of Prostate Cancer Patients with Biochemical Recurrence. J Nucl Med. 2018 Mar;59(3):434-441. doi: 10.2967/jnumed.117.202945. Epub 2017 Dec 14. PMID 29242398